CLINICAL TRIAL: NCT03060460
Title: Randomized Evaluation of Traditional Versus Ultrasound Guided Insertion of Sheath Before Angiography or Angioplasty
Brief Title: Ultrasound Guided Insertion of Sheath Before Angiography or Angioplasty
Acronym: ACCESS-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Christian Juhl Terkelsen (Other)
Responsible Party: Sponsor-Investigator, Christian Juhl Terkelsen, Associate professor, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: ACCESS-II
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Radial; Angioplasty; Angiography; Ultrasound; Randomized

STUDY DESIGN:
Intervention Model Description: historical control cohort (Group A) and then a randomized prospective study (Group B and C).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound arm - Randomized group (Experimental): Ultrasound guided sheath insertion
  Interventions: Diagnostic Test: Ultrasound guided sheath insertion
- Conventional arm - Randomized group (No Intervention): Conventional arm during randomized phase
- Historical control group (No Intervention): Conventional arm, non-randomization phase

INTERVENTIONS:
Diagnostic Test: Ultrasound guided sheath insertion — ultrasound is used routinely for sheath insertion
  Arms: Ultrasound arm - Randomized group

SUMMARY:
The study evaluates whether routine use of ultrasound for sheath insertion during radial or femoral angiography or angioplasty has any impact on: number of punctures, patient discomfort, procedural length, successfull procedure or ideal vessel puncture.

DETAILED DESCRIPTION:
A randomised study with an historical control group.

Initially data on prespecified endpoints are collected for an historical control group of 200 patients (100 radial and 100 femoral procedures). Hereafter 400 patients are randomized to ultrasound guided or conventional sheath insertion (200 radial and 200 femoral procedures).

Only high-volume physicians who have passed a ultrasound course are allowed to include patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for angiography or angioplasty in whom both radial and femoral access is possible

Exclusion Criteria:

* Abnormal pulse oxymetry test
* If severe lower-extremity calcification is known to exclude femoral access

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
number of puncture attempts | during the procedure
  Number of attempts to puncture the vessel as evaluated by the physician and by go-pro camera recordings
time of procedure | during the procedure
  time from administration of analgetics to removal of the sheath
Placement of sheath | during the procedure
  Distance from proc.styloideus radius (radial procedure) or proximal part of caput femoris (femoral procedure) to vessel puncture site evaluated by angiography
Pain during sheath insertion and during the procedure | during the procedure
  Pain according to numerical rating scale during sheath insertion and during the procedure
Successfull procedure | during the procedure
  Proportion of patients where the procedure is completed according to prespecified access route (no conversion to femoral access if radial planned, and no conversion to radial access if femoral planned)

SECONDARY OUTCOMES:
Use of analgetics | during the procedure
  Cummulated dose of analgetics during the procedure
Use of sedatives | during the procedure
  Cummulated dose of sedatives during the procedure
Use of calcium blocker | during the procedure
  Cummulated dose of calcium blocker during the procedure
Radial artery patency | during the procedure
  Patency according to reverse Barbeau test at time of sheath removal

CONTACTS AND LOCATIONS:
Overall Officials: erik sloth, professor, Study Chair — Department of anaestesiology, Aarhus University Hospital, DK-8200 Aarhus N
Locations (1):
- Department of cardiology, Aarhus University Hospital in Skejby, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Anonymous data can be shared